CLINICAL TRIAL: NCT01808963
Title: Evaluation of Respiratory Heat Loss as a Physiologic Patient Monitor for Acute Care Medicine
Brief Title: Evaluation of Respiratory Heast Loss as a Physiologic Patient Monitor for Acute Care Medicine
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 389048
Record Dates: First submitted 2013-03-07; First posted 2013-03-12 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Heat Loss
Keywords: Enthalpy; Physiologic Monitors; Critical Care Medicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the utility of respiratory heat loss measurements as a physiologic monitor.

DETAILED DESCRIPTION:
Respiratory Heat Loss Measured in Joules Per Minute

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical procedures.

Exclusion Criteria:

* Severe pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing elective surgery requiring arterial pressure monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal W Fleming, M.D., Ph.D, Principal Investigator — Director, Cardiovascular and Thoracic Anesthesiology
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 12/19/12 through 5/31/13 in the UCDMC Peri-operative Suite.
Groups:
- Study Group: Patients undergoing elective surgery requiring endotracheal intubation for anesthesia.
Period: Overall Study
Arm/Group | Study Group
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Respiratory Heat Loss Measured in Joules Per Minute
Arm/Group | Study Group
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Respiratory Heat Loss as a Physiologic Patient Monitor for Acute Care Medicine
Description: Respired gas heat content
Time Frame: 1 year.
Measure: Mean (Standard Deviation); unit: Joules per minute
Groups:
- Study Group: Joules per minute
Arm/Group | Study Group
Number analyzed (Participants) | 13
Joules per minute | 29.7 (15.6)

ADVERSE EVENTS:
Time Frame: 9 Months
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No